CLINICAL TRIAL: NCT00568204
Title: Proof of Concept of MEXYN-A
Brief Title: Study of Effectiveness of Mexyn-A
Acronym: Mexyn-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evangelical Synod Medical Centre (Other)
Responsible Party: Dr Ihab Akhnoukh M.D., Evangelical Synod Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EvangelicalSynodMC
Record Dates: First submitted 2007-11-30; First posted 2007-12-05 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Pruritus
Keywords: pruritus, itching, mexyn-a, clearitch, magicool-plus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Mexyn-A
  Interventions: Device: Mexyn-A

INTERVENTIONS:
Device: Mexyn-A — Atomised topical self-chilled pressurised spray
  Other Names: Clearitch, Itcharret, itchclear, Magicool-Plus

SUMMARY:
Atomised Methoxymethane-in-Aqua (MEXYN-A) a new topical self-chilled, non-steroidal, non-flammable, pressurised spray which embodies in one simultaneous application, most of the currently recognised and effective chemical, mechanical and thermal anti-pruritic therapies and hydrotherapy.

DETAILED DESCRIPTION:
The primary clinical endpoint was to establish MEXYN-A efficacy and safety in abolishing or reducing pruritus related to cutaneous diseases, insect bites and poison ivy, within few seconds of the application. The secondary endpoint was to measure the itch free period as a result of the new intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from severe itching due to : Atopic Dermatitis, contact dermatitis, psoriasis, urticaria, xerosis, prickly heat, genital pruritus, chicken pox, aquagenic pruritus, lichen planus, poison ivey, insect bites.
* Past experience with the use of at least one conventional medication for pruritus or conventional medication for the same disorder patients suffered.

Exclusion Criteria:

* Patients who have taken any anti-pruritic drug during the month prior to participation.
* Patients who have taken drugs for any reason for 2 days prior to participating in the study.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2002-03; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Treating Pruritus | three days

SECONDARY OUTCOMES:
measuring itch-free period after applying the new treatment, effect on sleep disturbance | three days

CONTACTS AND LOCATIONS:
Overall Officials: Ihab Akhnoukh, Principal Investigator — Evangelical Synod Medical Centre; Ashraf Khella, Study Director — Harpur Memorial Hospital
Locations (1):
- Evangelical Synod Medical Centre, Cairo, Cairo Governorate, Egypt